CLINICAL TRIAL: NCT02001025
Title: Performance of Bioabsorbable Vascular Scaffolds (Absorb) Compared to Xience Stents - an Optical Coherence Tomography Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rudolf Berger (Other)
Responsible Party: Sponsor-Investigator, Rudolf Berger, Associate Professor, Medical University of Vienna
Organization: Medical University of Vienna (Other)
Other Study IDs: Absorb/Xience 01
Record Dates: First submitted 2013-11-27; First posted 2013-12-04 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2013-11

CONDITIONS: Bioresorbable Scaffolds
Keywords: coronary vessels; coronary stenosis; percutaneous transluminal angioplasty; stents; drug-eluting stents; bioresorbable scaffolds; optical coherence tomography
MeSH Terms: conditions — Coronary Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Absorb scaffold: Bioresorbable vascular scaffold implanted in coronary arteries, which are completely resorbed over a period of approximately two years
  Interventions: Device: Absorb scaffold
- Xience stent: Second generation drug-eluting stent to treat coronary artery lesions
  Interventions: Device: Xience stent

INTERVENTIONS:
Device: Absorb scaffold
  Groups: Absorb scaffold
Device: Xience stent
  Groups: Xience stent

SUMMARY:
The biodegradable ABSORB scaffold is characterized by a greater strut thickness, but it has a greater flexibility compared to the XIENCE stent. Due to its fragility the inflating pressure of the ABSORB scaffold is limited and suitable lesions have to be well prepared. This study assesses the incidence of malapposed stent-struts, and the frequency of stent-underexpansion and edge dissection after ABSORB implantation compared to the XIENCE stent.

ELIGIBILITY:
Inclusion Criteria for implanting an Absorb scaffold:

* age < 55 years OR
* lesion length > 24mm OR
* multiple lesions to be treated

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with coronary artery disease
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2013-11; Primary Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
adverse post-stenting results | 1 year
  Malapposition, underexpansion and edge dissections assessed with Optical Coherence Tomography (OCT)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Vienna, Austria